CLINICAL TRIAL: NCT05404334
Title: Clinico-pathological Study of Androgen Receptor Expression in Breast Cancer With or Without BRCA Mutation
Brief Title: of Androgen Receptor Expression in Breast Cancer With or Without BRCA Mutation
Status: Completed | Type: Observational
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Banaras Hindu University
Other Study IDs: BRAR1
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin embedded blocks containing tumor and DNA will be retained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer: Patients with histologically proven breast cancer
  Interventions: Diagnostic Test: Androgen receptor status and BRCA mutation
- Benign breast disease: Patients with benign breast diseases undergoing surgical resection
  Interventions: Diagnostic Test: Androgen receptor status and BRCA mutation

INTERVENTIONS:
Diagnostic Test: Androgen receptor status and BRCA mutation — Androgen receptor status by IHC and germ line BRCA mutation

SUMMARY:
Androgen Receptor is extensively expressed in BRCA and its role in the disease may differ depending upon molecular subtypes and stages. Androgen Receptor (AR) may act as an antagonist of estrogen receptor α (ERα), in ERα induced effect, whereas in the absence of estrogens, AR may act as an agonist, of ERα- promoting tumor. Thus, depending on the BRCA micro-environment, both agonists and antagonists of the AR have been suggested for therapeutic approaches.

DETAILED DESCRIPTION:
The rate of AR positivity in breast cancer is about 60% to 80%. Biologically the AR pathway has cross talk with several other key signaling pathway, including the PI3K/Akt/mTOR and MAPK Pathways, and with other receptor, including estrogen receptor and human epidermal growth factor receptor-2. In clinical trials in patients with breast cancer, AR targeted therapies such as AR agonists, AR antagonists, PARP inhibitors, and PI3K inhibitors have shown promising results. The use of AR targeted therapies in conjunction with other agent has been investigated for overcoming resistance to AR focused treatments. Thus, the value of AR positivity as a prognostic marker has not been identified. Several retrospective clinical studies have shown that AR might be a prognostic or predictive factor in breast cancer. BRCA1 mutation accounts for the progress of hereditary breast cancers and is in connection with unique clinicopathological characteristics compared with sporadic breast cancers. The database is still evolving and newer mutation and their significance is being found every day. Also, there were several limitations to these previous studies. First, the cut-off for AR positivity was arbitrary. In most of the studies, the cut-off points were 1% or 10% and weren't enough to predict carcinoma survival. Moreover, quite 90% of the studies were conducted in non-Asian regions. Most of the studies involving Asian patients studied the prognostic role of AR in TNBC patients, with inconclusive results. There are only a few studies from Indian continents and none has correlated the AR expression with BRCA.

After the written inform consent in case of fresh recruitment the blood will be collected and tissue blocks will be obtained, use of already available blocks of patients who earlier participated in another study is also proposed.

(a) Samples will be stored for DNA study and will be frozen in liquid nitrogen and stored at -80 °C until further processing.

(samples will store in 10% formalin at room temperature (RT) for Immunohistochemistry

ELIGIBILITY:
Inclusion Criteria:

* Histology proven cases of breast cancer

Exclusion Criteria:

* Patients with prior treatment
* Pregnant and lactating women

Ages: 18 Years to 99 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer
Study Population: Patients with breast cancer and benign breast diseases
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Receptor expression | 6 months
  Androgen receptor expression and its correlation with molecular subtypes of breast cancer
BRCA1 and BRCA2 mutations | 6 months
  BRCA mutations and its correlation with molecular subtypes of breast cancer

SECONDARY OUTCOMES:
AR and BRCA | 6 months
  Correlation of Androgen receptor expression with BRCA mutation

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, MS, PhD, Principal Investigator — Banaras Hindu University
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months
Access Criteria: on request

REFERENCES:
- [Background] Anand A, Singh KR, Kumar S, Husain N, Kushwaha JK, Sonkar AA. Androgen Receptor Expression in an Indian Breast Cancer Cohort with Relation to Molecular Subtypes and Response to Neoadjuvant Chemotherapy - a Prospective Clinical Study. Breast Care (Basel). 2017 Jul;12(3):160-164. doi: 10.1159/000458433. Epub 2017 Jun 16. PMID 28785183
- [Background] Vidula N, Yau C, Wolf D, Rugo HS. Androgen receptor gene expression in primary breast cancer. NPJ Breast Cancer. 2019 Dec 10;5:47. doi: 10.1038/s41523-019-0142-6. eCollection 2019. PMID 31840050
- [Background] Zhang L, Fang C, Xu X, Li A, Cai Q, Long X. Androgen receptor, EGFR, and BRCA1 as biomarkers in triple-negative breast cancer: a meta-analysis. Biomed Res Int. 2015;2015:357485. doi: 10.1155/2015/357485. Epub 2015 Jan 28. PMID 25695063